CLINICAL TRIAL: NCT07092748
Title: A Phase I Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of HS387 in Subjects With Advanced Solid Tumors
Brief Title: A Phase Ia/ Ib Study of HS387 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS387-I-01
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS387 group (Experimental)
  Interventions: Drug: HS387

INTERVENTIONS:
Drug: HS387 — HS387 tablets will be given orally

SUMMARY:
This is a Phase Ia/Ib, dose escalation and dose expansion study to evaluate the safety, tolerability, PK, and preliminary efficacy of HS387 in subjects with advanced solid tumors. It includes two parts: the dose escalation study (Phase Ia) and the dose expansion study (Phase Ib)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

  1. Men or women ≥18 years old and ≤75 years old.
  2. Subjects with advanced solid tumors who have failed or are intolerant to standard treatment, or have no standard therapy.
  3. Survival expectation is ≥ 3 months.
  4. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
  5. Phase Ⅰa: Subjects with advanced solid tumors have at least one evaluable lesion according to RECIST 1.1. Phase Ⅰb: Subjects with advanced solid tumors have at least one measurable lesion according to RECIST 1.1.
  6. Subjects with adequate organ function at the time of screening.
  7. Serum pregnancy test (for female of childbearing potential) negative prior to first dosing of study treatment. Male and female subjects of childbearing potential must agree to use effective methods of contraception throughout the study and for 3 months after the last dose of the investigational product.

     Exclusion Criteria:
* Subjects will be excluded if they meet any of the following criteria:

  1. Has received other investigational drugs or treatments not yet approved for marketing within 4 weeks prior to the first administration.
  2. Has active infection.
  3. Has meningeal metastases or symptomatic central nervous system (CNS) metastases.
  4. Significant impairment of oral drug absorption.
  5. Has interstitial lung disease.
  6. Pregnant or lactating women.
  7. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
  8. Has a major surgical procedure within 4 weeks prior to the first administration.
  9. Has a treatment history of KIF18A inhibitor.
  10. In the opinion of the Investigator, there are other factors that the subject is unsuitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting Adverse Events (AEs) or Serious Adverse Events (SAEs) | 2 years
  Adverse events (AE), serious adverse events (SAE), and severity of AE using the NCI-CTCAE version 5.0
Dose-limiting Toxicities Incidence Count Among Study Participant | 2 years
  DLT refers to Dose-Limiting Toxicity. It is defined as a side effect or adverse reaction of a drug or treatment that is severe enough to prevent an increase in dosage. Identifying DLT is crucial in clinical trials for determining the maximum tolerated dose (MTD) of a new drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer hospital, Hangzhou, Zhejiang, China